CLINICAL TRIAL: NCT05004844
Title: Mitochondrial Dysfunction in Trauma-related Coagulopathy - Is There Causality? - Study Protocol for a Prospective Observational Study
Brief Title: Mitochondrial Dysfunction in Trauma-related Coagulopathy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Petra Hartmann MD Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Petra Hartmann MD Ph.D., Associate Professor, Szeged University
Organization: Szeged University (Other)
Other Study IDs: 5500/2021-SZTE
Record Dates: First submitted 2021-08-06; First posted 2021-08-13 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-09

CONDITIONS: Trauma Induced Coagulopathy
Keywords: blood coagulation disorders; wounds and injuries; hemorrhage; mitochondria; blood platelet disorders; thrombelastography; coagulopathy, trauma induced
MeSH Terms: conditions — Blood Coagulation Disorders; Wounds and Injuries; Hemorrhage; Blood Platelet Disorders; Hemostatic Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Viscoelastic assays and aggregometry tests — Viscoelastic assays and aggregometry tests performed with ROTEM will allow us to characterize the clot forming abilities and platelet functions of our patients. ROTEM is used routinely for aiding clinicians in choosing the appropriate blood products for patients ROTEM requires samples of whole blood in an amount that does not entail additional burden or risk for patients. In our study, viscoelastic assays and aggregometry will be performed upon arrival, and 24-,48-,72-hours post-admission.

SUMMARY:
Bleeding control often poses a great challenge for clinicians due to trauma-induced blood clotting disorder (TIC), a condition that is present in one-third of bleeding trauma patients. As platelets are considered as central mediators in TIC, the understanding of mitochondria-mediated processes in thrombocytes may disclose new therapeutic targets in the management of severely injured patients. The investigators hypothesize that mitochondrial dysfunction occurs in the platelets of trauma patients with TIC. The investigators intend to quantitatively characterize the derangements of mitochondrial functions in TIC; and assess the relation between mitochondrial respiration and clinical markers of platelet function

DETAILED DESCRIPTION:
Hemorrhage control often poses a great challenge for clinicians due to trauma-induced coagulopathy (TIC), a condition that is present in one-third of bleeding trauma patients. As platelets are considered as central mediators in TIC, the understanding of mitochondria-mediated processes in thrombocytes may disclose new therapeutic targets in the management of severely injured patients. The investigators hypothesize that mitochondrial dysfunction occurs in the platelets of trauma patients with TIC. The investigators intend to quantitatively characterize the derangements of mitochondrial functions in TIC; and assess the relation between mitochondrial respiration and clinical markers of platelet function measured with aggregometry, viscoelastic tests and conventional laboratory analysis.

ELIGIBILITY:
Inclusion Criteria:

* Trauma patients
* Injury Severity Score (ISS) 16 or greater,
* age of 18 years or greater,
* hemorrhage confirmed with extended focused assessment with sonography in trauma (eFAST) or computer tomography (CT)

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Severely injured trauma patients with hemorrhage
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-10-31 (Estimated); Primary Completion 2022-10-31 (Estimated); Study Completion 2023-01-31 (Estimated)

PRIMARY OUTCOMES:
Association between mitochondrial functions and aggregation capacity of platelets | 72 hours
  The association between the results of high-resolution respirometry (The activity of respiratory complexes, the ATP synthase activity (OxPhos), the electron transport chain capacity and coupling of mitochondria) and numerical parameters of ROTEM aggregometry (AUC, MS and A6 in TRAPTEM) at 0, 24, 48, and 72 hours post-admission will constitute our primary outcome.

SECONDARY OUTCOMES:
Association between platelet mitochondrial functions and clot formation ability | 72 hours
  The association between the results of high-resolution respirometry (The activity of respiratory complexes, the ATP synthase activity (OxPhos), the electron transport chain capacity and coupling of mitochondria) and results of viscoelastic assays (CT, CFT, α-angle, A10, MCF, LI30 and ML in INTEM, EXTEM, APTEM, FIBTEM) at 0, 24, 48, and 72 hours post-admission will serve as secondary outcome.
Association between platelet mitochondrial functions and conventional laboratory markers of hemostasis | 72 hours
  The association between the results of high-resolution respirometry (The activity of respiratory complexes, the ATP synthase activity (OxPhos), the electron transport chain capacity and coupling of mitochondria) and conventional markers of hemostasis (prothrombin time (PT), International Normalized Ratio (INR)) at 0, 24, 48, and 72 hours post-admission will serve as secondary outcome.
Relation between platelet mitochondrial functions and mortality | 72 hours
  The association between the results of high-resolution respirometry (The activity of respiratory complexes, the ATP synthase activity (OxPhos), the electron transport chain capacity and coupling of mitochondria) and 72-hour mortality will serve as secondary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Endre Prof. Dr. Varga, M.D,Ph.D,DSc, Study Director — Department of Traumatology, University of Szeged; Petra Dr. Hartmann, M.D., Ph.D., Principal Investigator — Department of Traumatology, University of Szeged
Locations (1):
- Department of Traumatology, University of Szeged, Szeged, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Moore EE, Moore HB, Kornblith LZ, Neal MD, Hoffman M, Mutch NJ, Schochl H, Hunt BJ, Sauaia A. Trauma-induced coagulopathy. Nat Rev Dis Primers. 2021 Apr 29;7(1):30. doi: 10.1038/s41572-021-00264-3. PMID 33927200
- [Background] Barile CJ, Herrmann PC, Tyvoll DA, Collman JP, Decreau RA, Bull BS. Inhibiting platelet-stimulated blood coagulation by inhibition of mitochondrial respiration. Proc Natl Acad Sci U S A. 2012 Feb 14;109(7):2539-43. doi: 10.1073/pnas.1120645109. Epub 2012 Jan 30. PMID 22308457
- [Background] Kornblith LZ, Moore HB, Cohen MJ. Trauma-induced coagulopathy: The past, present, and future. J Thromb Haemost. 2019 Jun;17(6):852-862. doi: 10.1111/jth.14450. Epub 2019 May 13. PMID 30985957
- [Background] Kutcher ME, Redick BJ, McCreery RC, Crane IM, Greenberg MD, Cachola LM, Nelson MF, Cohen MJ. Characterization of platelet dysfunction after trauma. J Trauma Acute Care Surg. 2012 Jul;73(1):13-9. doi: 10.1097/TA.0b013e318256deab. PMID 22743367
- [Derived] Javor P, Rarosi F, Horvath T, Torok L, Hartmann P. Mitochondrial Dysfunction in Trauma-Related Coagulopathy: Is There Causality? Study Protocol for a Prospective Observational Study. Eur Surg Res. 2023;64(2):304-309. doi: 10.1159/000521670. Epub 2021 Dec 24. PMID 34954696